CLINICAL TRIAL: NCT03262428
Title: Collaborative Self-Management Support in Chronic Conditions: a Qualitative Study of Patients', Caregivers' and Health Care Professionals' Views and Experiences of Integrated Care in Asthma, Breast Cancer and Stroke
Brief Title: Collaborative Self-Management Support in Chronic Conditions - Qualitative Study
Acronym: CoSMaS-ql
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0480
Record Dates: First submitted 2017-08-24; First posted 2017-08-25 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Asthma; Breast Cancer; Stroke
MeSH Terms: conditions — Asthma; Breast Neoplasms; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: Patients with asthma, breast cancer, and stroke living in the Rhône Alpes region
  Interventions: Other: Semi-structured interviews
- Caregivers: Caregivers of patients with asthma, breast cancer, and stroke living in the Rhône Alpes region
  Interventions: Other: Semi-structured interviews
- Health care professionals: Health care professionals involved in the care of patients with asthma, breast cancer, and stroke living in the Rhône Alpes region
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — Patients, caregivers and health care professionals involved in self-management support will be sought via patient organizations and professional organizations in the region. Study information materials will be provided to these organizations for dissemination to their members, providing also contact details of the study team for interested individuals to register their interest and provide basic eligibility and screening information. Selected participants will be invited to take part in a face-to-face or telephone interview about (supporting) self-management. Data collection will consist of semi-structured interviews conducted either face-to-face or by telephone.

SUMMARY:
The management of chronic conditions is a challenge for health systems worldwide, particularly in the context of an aging population, and requires urgent improvement of health services. Integrated care and patient empowerment represent promising solutions: offering tailored self-management support in a collaborative framework led to good results in several clinical contexts. Yet, large scale implementation remains a challenge. An important limitation of existing solutions is a lack of utilization of behavioural and communication theory for identifying the dynamics of pluridisciplinary collaboration and the interactive effects of the activities performed by several actors involved in self-management support in a given chronic condition. A second limitation is not involving all relevant actors in the development of health service improvement solutions, which leads to limited programme adoption and sustainability in routine care.

This study is part of a project that proposes to address these limitations and develop and interdisciplinary model of collaborative care in the self-management of chronic conditions (CoSMaS) that adopts a community-based participative approach. CoSMaS-ql is a qualitative study that will consist of semi-structured interviews with several types of stakeholders: patients, caregivers, and health care professionals of different specialties (e.g. general practitioners, nurses, specialist consultants, pharmacists). The main objective of the study is to explore the experiences and of patients, caregivers, and HCPs on how self-management support is currently delivered in asthma, cancer and stroke (content, communication, organisation of care), their needs related to self-management support provision, and envisaged solutions for improving current practice. Three different chronic conditions will be targeted: asthma, breast cancer and stroke. The qualitative data will be analysed via grounded-theory and template analysis. It will inform the development of a theoretical model of collaborative self-management support in chronic conditions. It will also result in three profiles describing 'real' versus 'ideal' care processes, which will represent needs assessment stages for future health services improvement interventions in the three conditions.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* having (had) one of the health conditions targeted.
* age >18 years (in order to have had the opportunity to achieve full transition from parent/caregiver-managed to self-managed care),
* at least 1 year since diagnosis (in order to have had sufficient time to experience adjustments to their condition on the long term), and
* at least 1 consultation with an HCP of any specialty in the past year (in order to ensure minimum 1 recent experience of care they could reflect on).

Exclusion Criteria:

* unable to communicate in French
* level of severity of health condition or comorbidities making participation in the study too burdensome

CAREGIVERS:

Inclusion Criteria:

- nominated by a participating patients as principal caregiver

Exclusion Criteria:

- none

HEALTH CARE PROFESSIONALS :

Inclusion Criteria:

- at least 1 year of experience working in one of the 3 chronic conditions targeted (irrespective of the number of patients consulted)

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be patients, caregivers and health care professionals in the Rhône Alpes region involved in self-management support in cancer, asthma or stroke.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2018-04-14 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Experiences and views of patients, caregivers, and health care professionals involved in the long-term management of asthma, cancer and stroke about real and ideal practices in collaborative self-management support. | About 60 minutes
  Interviews will be semi-structured and follow a topic guide designed to explore participants' goals, behaviours and determinants, perceptions of others' goals and behaviours, communication processes, tools used in self-management, support, and communication, and their vision on optimal processes and ways to implement them. Caregivers will be interviewed separately on their experiences of caregiving and self-management support by HCPs. HCPs will be interviewed regarding their experiences of providing care in one or more of the 3 chronic conditions (depending on their experience and time constraints) and their thoughts on collaborating with other professionals and solutions for integrated care and ensuring continuity of care.

CONTACTS AND LOCATIONS:
Locations (1):
- EA 7425 HESPER - Health Services and Performance Research, Université Claude Bernard Lyon 1, Lyon, France

IPD SHARING:
Plan to Share IPD: No